CLINICAL TRIAL: NCT03894995
Title: Optimizing Windows to Improve Ventilation in Dhaka Slums
Brief Title: Optimizing Ventilation to Improve Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Johns Hopkins University (Other); University at Buffalo (Other)
Responsible Party: Principal Investigator, Stephen P Luby, Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 46212
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Pollution; Exposure
Keywords: Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1. Focus group discussions on ventilation preferences (No Intervention): Participant's perceived benefits/detriments of having ventilation options in the household and their opinions on the behavior change material developed to encourage increased household ventilation will be explored using 6-9 focus group discussions with 10-12 participants each.
- Part 2. PM 2.5 pilot (No Intervention): Indoor, outdoor, and personal particulate matter concentrations among ten mother-child pairs and their homes will be monitored.
- Part 3. Intervention (Experimental): Households will participate in a baseline survey and a Beck-DeGroot-Marshak auction to establish willingness-to-pay for ventilation. If the household wins, or if it is decided to install ventilation in all intervention households, the household will receive installation of a ventilating mechanism.
  Interventions: Other: Installation of ventilation
- Part 3. Control (No Intervention): For 12 month after intervention, the air exchange rate will be measured in all control households.
- Part 4. Spillover (No Intervention): Households that neighbor enrolled study households will be surveyed and asked whether they, on their own, chose to install a window. If they did install a window, they will be asked how much they paid.

INTERVENTIONS:
Other: Installation of ventilation — The intervention is installation of a ventilating structure, in this case a window in the house roof.
  Arms: Part 3. Intervention

SUMMARY:
Our overall goal is to optimize preferred, ventilating windows/apertures/vents in low-income neighborhoods of Dhaka, Bangladesh. We will:

I. Collect baseline data on housing types and finalize windows/vents protoypes.

II. Measure the impact of improved ventilation on air exchange rates in houses in low-income neighborhoods of Dhaka and characterize the current and potential market for windows/vents in households in low-income neighborhoods of Dhaka, Bangladesh.

III. Understand recipients' (tenants and landords) perceived benefits of installed window/vent designs and difficulties faced with adoption of each design

ELIGIBILITY:
Inclusion Criteria:

* 1) lack cross-ventilation at the time of enrollment
* 2) have obtained landlord permission to make adjustments to their dwelling,
* 3) have a free roof where a window can be installed

Exclusion Criteria:

* 1) Household reports receiving dust from nearby machine that pulverizes materials for making roads

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Household air exchange rate - spring (Part 3) | 50 minutes
  Repeated household measurements of effective point ventilation to approximate air exchange rates in both treatment and control households will be obtained. Air exchange rates will be reported as air changes per hour for the home as well as liters of air per cubic meter per second per person.
Household air exchange rate - summer (Part 3) | 50 minutes
  Repeated household measurements of effective point ventilation to approximate air exchange rates in both treatment and control households will be obtained. Air exchange rates will be reported as air changes per hour for the home as well as liters of air per cubic meter per second per person.
Household air exchange rate - fall (Part 3) | 50 minutes
  Repeated household measurements of effective point ventilation to approximate air exchange rates in both treatment and control households will be obtained. Air exchange rates will be reported as air changes per hour for the home as well as liters of air per cubic meter per second per person.
Household air exchange rate - winter (Part 3) | 50 minutes
  Repeated household measurements of effective point ventilation to approximate air exchange rates in both treatment and control households will be obtained. Air exchange rates will be reported as air changes per hour for the home as well as liters of air per cubic meter per second per person.
Number of households that adopt the intervention (Part 3) | 20 minutes
  Takeup of the intervention will be defined by whether a household had a ventilation design installed, either by winning the BDM auction paying the full price or by accepting a free installation after previously losing the BDM auction.
Revealed willingness-to-pay for ventilation (Part 3) | 20 minutes
  We will obtain stated willingness-to-pay for the ventilation designs through the BDM auction mechanism, which will be used to trace out a demand curve for ventilation, plotting the number of households that are willing to pay for a window agaist their stated price.
Concentration of radon gas in house (Part 3) | 7 days
  We will assess the concentration gas in a subset of study households.
Concentration of indoor particulate matter 2.5 (Part 3) | 48 hours for normal tests; 72 hours for quality control tests.
  We will determine the indoor PM2.5 levels in study households, as well as the number of hours with indoor PM2.5 exceeding 50 and 100 µg/m3 during the observation period. A subset of households will have longer tests for quality control.
Concentration of indoor particulate matter 2.5 (Part 2) | up to 5 hours
  We will determine the indoor PM2.5 levels in study households, as well as the number of hours with indoor PM2.5 exceeding 50 and 100 µg/m3 during the observation period.
Concentration of outdoor particulate matter 2.5 (Part 2) | up to 5 hours
  We will determine the outdoor PM2.5 levels near the study households.
Personal exposure to particulate matter 2.5 - mother (Part 2) | up to 5 hours
  We will determine the PM2.5 levels near the mother using a monitor worn on her body.
Personal exposure to particulate matter 2.5 - child (Part 2) | up to 5 hours
  We will determine the PM2.5 levels near the child using a monitor worn on her body.
Number of non-study, neighboring households that adopt the intervention and their willingness to pay (Part 4) | 15 minutes
  We will survey households that neighbor enrolled study households to ask if they have installed a window on their own since the enrollment for the randomized control trial. If they did install a window, we will ask how much they paid.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Luby, Dr., Principal Investigator — Stanford University
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No